CLINICAL TRIAL: NCT03382873
Title: Impact of Augmented Care at the Worksite for Diabetes Prevention
Brief Title: Augmented Care at Worksite for Diabetes Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Carla Miller, Professor (current affiliation at Indiana University), Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK112930-01A1 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: PreDiabetes
Keywords: Hyperglycemia; Obese; Overweight
MeSH Terms: conditions — Prediabetic State; Hyperglycemia; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: The proposed translational study applied an innovative experimental approach, an adaptive design, to optimize treatment for weight loss and weight loss maintenance in individuals with prediabetes. All participants initiated a standard lifestyle intervention to promote weight loss. Those who did not achieve >2.5% weight loss during the first month of the intervention were stratified to augmented care to enhance weight loss during the intensive intervention phase. Following the intensive phase, participants were randomly assigned to either the standard intervention or the enhanced intervention for the maintenance study phase. By randomly assigning participants to either the standard maintenance phase of the intervention or the innovative maintenance phase of the intervention following the initial core phase, the impact of extended training in self-regulation for weight loss maintenance was evaluated.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Lifestyle Balance (GLB) (Active Comparator): Standard lifestyle intervention to promote weight loss
  Interventions: Behavioral: Group Lifestyle Balance (GLB)
- Group Lifestyle Balance Plus (GLB+) (Experimental): Augmented lifestyle intervention for early slow responders
  Interventions: Behavioral: Group Lifestyle Balance Plus (GLB+)

INTERVENTIONS:
Behavioral: Group Lifestyle Balance (GLB) — The intervention included the following key features: group-based sessions led by a lifestyle coach; a structured, state-of-the-art, 16-session core-curriculum that emphasized behavioral self-management strategies for weight loss and physical activity; 8-months of extended care with bimonthly or monthly sessions; self-monitoring of diet and physical activity.
  Arms: Group Lifestyle Balance (GLB)
Behavioral: Group Lifestyle Balance Plus (GLB+) — The GLB+ intervention arm included participants who did not achieve the targeted percent weight loss by week 5 and incorporated enhanced training in values clarification, mindful decision making, planning, and problem solving. GLB+ included the same number of group-based sessions as GLB.
  Arms: Group Lifestyle Balance Plus (GLB+)

SUMMARY:
The purpose of the study was to evaluate the impact of augmented care at the worksite through a lifestyle intervention for diabetes prevention among employees with prediabetes who were slower to respond to a standard diabetes prevention intervention.

DETAILED DESCRIPTION:
Employees at the Ohio State University (OSU) with prediabetes participated in a standard lifestyle intervention (Group Lifestyle Balance) for diabetes prevention. Participants who did not achieve >2.5% weight loss at week 5 of the intervention were stratified to the augmented intervention (Group Lifestyle Balance Plus) at week 5. The impact of the augmented intervention compared to the standard intervention was determined at 4, 12 and 18 months from baseline to determine if implementing early enhanced training helped participants achieve and maintain weight loss similar to those who received the standard intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Benefits-eligible Ohio State University (OSU) employee
2. Intend to be employed by OSU through the length of the follow-up phase
3. Body mass index: >24 kg/m^2 non-Asians; >22 kg/m^2 Asians
4. Fasting blood glucose of 100-125 mg/dL or an A1c of 5.7-6.4%
5. Blood glucose of 110-199 (if non-fasting in previous 2 hours)

Exclusion Criteria:

1. Blood glucose level of ≥ 200 mg/dL
2. Conditions that would limit adoption of light/moderate physical activity (i.e., cardiac event, severe chronic obstructive pulmonary disease, advanced arthritis, poorly controlled hypertension)
3. Chronic use of medications that affect blood glucose levels (i.e., corticosteroids)
4. Concurrent participation in a structured weight loss program or counseling for bariatric surgery
5. Pregnant or breastfeeding
6. Score of ≥ 10 on the Patient Health Questionnaire-8 indicating moderate to severe depressive symptoms
7. Score of ≥ 27 on the Binge Eating Scale indicating the potential for binge eating
8. Unwilling to accept randomization
9. Planning to move from the area or changing employment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Miller, Ph.D., Principal Investigator — The Ohio State University (during study implementation)
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be released to other researchers using a data-sharing agreement that specifies that the data will be used only for research purposes and only by the specified individuals to whom the data are released. Documentation of Institutional Review Board approval for the proposed use must be provided in advance to the PI. The data must be either destroyed or returned to the PI after all analyses are completed.
Supporting Information: CSR
Time Frame: The data will be available following all analyses and publication of primary and secondary study results. The data will be available upon request.
Access Criteria: To be developed

REFERENCES:
- [Derived] Miller CK, Nagaraja HN, Cheavens JS, Fujita K, Lazarus SA, Brunette DS. Sex Differences in Early Weight Loss Success During a Diabetes Prevention Intervention. Am J Health Behav. 2023 Apr 30;47(2):337-348. doi: 10.5993/AJHB.47.2.13. PMID 37226352
- [Derived] Miller CK, King D, Nagaraja HN, Fujita K, Cheavens J, Focht BC. Impact of an augmented intervention on self-regulatory, dietary and physical activity outcomes in a diabetes prevention trial among adults with prediabetes. J Behav Med. 2023 Oct;46(5):770-780. doi: 10.1007/s10865-023-00406-w. Epub 2023 Mar 18. PMID 36933057
- [Derived] Miller CK, Nagaraja HN, Cheavens J, Fujita K, Lazarus S. Impact of a Novel Diabetes Prevention Intervention for Early Slow Weight Loss Responders Among Adults With Prediabetes: An Adaptive Trial. Diabetes Care. 2022 Oct 1;45(10):2452-2455. doi: 10.2337/dc22-0824. PMID 36041053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Employees from a Midwestern university with overweight or obesity and prediabetes were recruited from 2018-2021.
Pre-assignment Details: Participants completed 4 weeks of the standard Group Lifestyle Balance (GLB) intervention. Those who achieved >2.5% weight loss at week 5 remained in GLB at week 5. Those who achieved <2.5% weight loss at week 5 were stratified to the GLB Plus (GLB+) intervention at week 5. Participants were paired based on percent weight change at month 5. Each member in the pair was randomized to group at month 5 for the study duration. Thus, group sample sizes are different at month 5 compared to month 4.
Groups:
- Group Lifestyle Balance (GLB): Standard lifestyle intervention
- Group Lifestyle Balance Plus (GLB+): Augmented lifestyle intervention for slow responders
Period: Overall Study
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
Started | 86 | 122
Completed 4-months | 80 | 111
Randomized at 5-months | 94 | 96
Completed 12-months | 87 | 88
Completed 18-months | 55 | 60
Completed | 55 | 60
Not Completed | 31 | 62
Not completed — Lost to Follow-up | 9 | 10
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Visit not completed due to pandemic | 16 | 41

BASELINE CHARACTERISTICS:
Population: Excludes people who withdrew from the study following stratification to treatment group
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+) | Total
Number analyzed (Participants) | 80 | 111 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (10.0) | 51.5 (10.2) | 52.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 90 | 140
  Male | 30 | 21 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 79 | 105 | 184
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 18 | 23
  White | 70 | 81 | 151
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 2
Body weight [Least Squares Mean (Standard Deviation); unit: kg] | 102.6 (2.7) | 102.5 (2.3) | 102.5 (1.8)
Fasting glucose [Least Squares Mean (Standard Deviation); unit: mg/dL] | 109.24 (1.14) | 107.58 (0.99) | 108.1 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Percent Weight Change
Description: Change in weight as measured in light clothing and shoes removed
Time Frame: baseline and 4-months
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
Number analyzed (Participants) | 80 | 111
percent change | -8.13 (0.48) | -3.46 (0.31)
Statistical Analysis 1: Comparison: Group Lifestyle Balance (GLB) vs Group Lifestyle Balance Plus (GLB+); Test type: Superiority; p < 0.0001, ANOVA

2. Primary Outcome: Percent Weight Change
Description: Change in weight as measured in light clothing and shoes removed
Time Frame: baseline and 12-months
Population: Compares the change for the GLB/GLB intervention sequence to the GLB+/GLB+ intervention sequence (the primary comparison of interest at 12-months)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
Number analyzed (Participants) | 47 | 59
percent change | -9.55 (0.96) | -4.00 (1.05)
Statistical Analysis 1: Comparison: Group Lifestyle Balance (GLB) vs Group Lifestyle Balance Plus (GLB+); Compares the change for the GLB/GLB intervention sequence to the GLB+/GLB+ intervention sequence (the primary comparison of interest); Test type: Superiority; p = 0.0001, ANOVA; Intervention sequence and sex were used as independent predictors in the model

3. Primary Outcome: Percent Weight Change
Description: Change in weight as measured in light clothing and shoes removed
Time Frame: 12-months and 18-months
Population: Compares the GLB/GLB intervention sequence to the GLB+/GLB+ intervention sequence (the primary comparison of interest at 18-months for weight loss maintenance)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
Number analyzed (Participants) | 27 | 42
percent change | 2.22 (0.59) | 2.28 (0.56)
Statistical Analysis 1: Comparison: Group Lifestyle Balance (GLB) vs Group Lifestyle Balance Plus (GLB+); Comparison of the GLB/GLB intervention sequence to the GLB+/GLB+ intervention sequence (the primary comparison of interest); Test type: Superiority; p = 0.9476, ANOVA; Intervention sequence and sex used as independent predictors in the model

4. Secondary Outcome: Fasting Glucose
Description: Fasting glucose from a fingerstick sample
Time Frame: baseline and 4-months
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
Number analyzed (Participants) | 80 | 111
mg/dL | -7.01 (1.13) | -3.18 (0.98)
Statistical Analysis 1: Comparison: Group Lifestyle Balance (GLB) vs Group Lifestyle Balance Plus (GLB+); Test type: Superiority; p = 0.0112, ANOVA; Treatment group, time and their interaction were fixed effects and participants were random effects

5. Secondary Outcome: Fasting Glucose
Description: Fasting glucose from a fingerstick sample
Time Frame: baseline and 12-months
Population: Compares the GLB/GLB intervention sequence to GLB+/GLB+ intervention sequence (the primary comparison of interest at 12-months)
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
Number analyzed (Participants) | 47 | 59
mg/dL | -4.30 (1.57) | -4.04 (1.70)
Statistical Analysis 1: Comparison: Group Lifestyle Balance (GLB) vs Group Lifestyle Balance Plus (GLB+); Comparison of GLB/GLB intervention sequence to GLB+/GLB+ intervention sequence (the primary comparison of interest); Test type: Superiority; p = 0.9085, ANOVA; Intervention sequence and sex used as independent predictors in the model

6. Secondary Outcome: Fasting Glucose
Description: Fasting glucose from a fingerstick sample
Time Frame: 12-months and 18-months
Population: Compares the GLB/GLB intervention sequence to the GLB+/GLB+ intervention sequence (the primary comparison of interest at 18-months)
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
Number analyzed (Participants) | 27 | 42
mg/dL | -1.21 (2.28) | 2.71 (2.08)
Statistical Analysis 1: Comparison: Group Lifestyle Balance (GLB) vs Group Lifestyle Balance Plus (GLB+); Comparison between the GLB/GLB intervention sequence and the GLB+/GLB+ intervention sequence (the primary comparison of interest); Test type: Superiority; p = 0.2063, ANOVA; Intervention sequence and sex used as independent predictors in the model

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse events were collected at every participant contact using a standardized form.
Arm/Group | Group Lifestyle Balance (GLB) | Group Lifestyle Balance Plus (GLB+)
All-Cause Mortality (participants affected / at risk) | 0/86 | 1/122
Serious Adverse Events (participants affected / at risk) | 2/86 | 3/122
Other Adverse Events (participants affected / at risk) | 4/86 | 13/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Lifestyle Balance (GLB) (N=86) | Group Lifestyle Balance Plus (GLB+) (N=122)
Hamstring tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Arrythmia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Colon abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hand surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Lifestyle Balance (GLB) (N=86) | Group Lifestyle Balance Plus (GLB+) (N=122)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Knee or hip pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)

LIMITATIONS AND CAVEATS:
Four participant cohorts did not complete the 18-month visit due to pandemic-related restrictions during the SARS-CoV-2 pandemic. Thus, the 18-month outcomes include a smaller sample and should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT03382873/Prot_SAP_000.pdf